CLINICAL TRIAL: NCT02408952
Title: Screening for Youth Alcohol and Drug Use: A Study of Primary Care Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 11-07796
Record Dates: First submitted 2015-03-20; First posted 2015-04-06 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Substance Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Physicians, Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary Care Physician (Experimental): If the adolescent is identified at risk for substance use, the screening and brief intervention referral to treatment delivered is by the primary care physician
  Interventions: Behavioral: Primary Care Physician
- Behavioral Medicine Specialist (Experimental): If the adolescent is identified at risk for substance use, the screening and brief intervention referral to treatment delivered by the behavioral medicine specialist
  Interventions: Behavioral: Behavioral Medicine Specialist
- Usual Care (No Intervention): Care is administered as usual

INTERVENTIONS:
Behavioral: Primary Care Physician — The screening, brief intervention and referral to treatment is delivered by the Primary Care Physician
  Arms: Primary Care Physician
Behavioral: Behavioral Medicine Specialist — The screening, brief intervention and referral to treatment is delivered by the Behavioral Medicine Specialist.
  Arms: Behavioral Medicine Specialist

SUMMARY:
This study evaluates the implementation and effectiveness of two modalities of Screening, Brief Intervention and Referral to Treatment (SBIRT) to reduce adolescent alcohol and other drug (AOD) use in a large pediatrics clinic.

DETAILED DESCRIPTION:
Health systems have not implemented Screening, Brief Intervention and Referral to Treatment (SBIRT) for adolescents despite research demonstrating its effectiveness. Based on prior research that identified barriers to AOD screening for adolescents in pediatric Primary Care (PC) and a pilot study that found SBIRT was feasible, well-received and promoted referrals to and initiation of specialty treatment, the current research application proposes to randomize 45 Primary Care Physicians (PCPs) in the pediatrics clinic of a medical center within a large, managed care health system, Kaiser Permanente Northern California, to three arms - 1) Usual Care; 2) SBIRT delivered by PCPs; and 3) SBIRT delivered by Behavioral Medicine Specialists (BMS). The study objective is to compare the implementation, effectiveness and cost-effectiveness of SBIRT for adolescents in PC in the three study arms. Patients will complete evidence-based screening and AOD assessment measures which have been embedded in the health plan's electronic medical record (EMR). A mixed model will be used to compare implementation outcomes (rates of screening and identification, brief intervention, referral to Chemical Dependency treatment and treatment initiation), and effectiveness (patient outcomes of AOD use and abstinence) at 12 months. The model accounts for the intra-class correlations across patients within providers. Cost-effectiveness relative to implementation and patient outcomes will be examined. Barriers and facilitators of implementation, and feasibility via qualitative interviews with clinicians and administrators will be examined as well. The study is significant in that it examines issues that must be addressed to spur widespread adaptation of SBIRT. The proposed interventions are highly feasible in the current environment of health reform due to increased resources and training to Federally Qualified Health Centers and private health plans. It is innovative in using the EMR to change clinical practice and systematically integrate AOD in PC, and as a platform for collecting research data.

ELIGIBILITY:
There are two study populations as described below thus the large age limit range.

Inclusion Criteria:

* All adolescent primary care providers at the pediatric primary care clinic will be included.
* All adolescent patient electronic records, ages 12-18, at the pediatric primary care will be examined.

Exclusion Criteria:

* Any adolescent primary care providers not practicing at the pediatric primary care clinic research site will be excluded.
* Adolescents electronic records who are not part of the research site pediatric clinic will be excluded.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9084 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening rate | Initial screening rate - at index well-visit
  The proportion of patients who are screened with the Teen Well Check Questionnaire AOD use or Mood symptom questions, among all patients with Teen well-child visits.
Problem Identification rate | Initital problem identification rate - at index well-visit, following screening
  The proportion of patients screened who answer "yes" to AOD use or Mood symptoms in past 12 months and "yes" to at least one non-car CRAFFT question. (Being in a car with someone using AOD may not be related to child's problem, but to having a parent/other adult who has driven while drinking/using).
Assessment rate | Within 2 weeks following index well-visit date
  Proportion of patients screening positive for alcohol or other drug, or mental health risk, who are assessed further using the CRAFFT tool.
Brief Intervention rate | Within 14 days of assessment at index well visit
  The proportion of patients who receive an intervention within 14 days, among those who are identified with AOD risk (based on CRAFFT score). Documented in EHR by clinicians, using an ICD-9 Administrative V-code for substance use counseling or behavioral counseling.
Referral to specialty treatment rate | Within 6 months of index well-visit
  The proportion of patients who receive referrals to specialty behavioral health treatment, among those identified through the CRAFFT as needing such treatment. Documented in the EHR.

SECONDARY OUTCOMES:
Specialty Behavioral Health Treatment Initiation | Within 2 years post-intervention
  Defined as the percent referred, who have at least one specialty behavioral health visit among those identified with a behavioral health problem. Documented in the EHR.
Alcohol and other drug use | Use in past 6 months, at 1 and 2 years post-intervention
  Alcohol and drug use: The items in the EHR measure past 30-day and 6-month use of alcohol, marijuana and other drugs and tobacco, including days of use, quantity consumed (any, 3+ and 5+ drinks), and days of binge drinking (3+ and 5+).
Substance Use-related outcomes | in past 6 months, at 1 and 2 years post-intervention
  AOD-related legal, school, and family problems: The EHR questions also include measures from the Comprehensive Adolescent Severity Inventory (CASI),148 a semi-structured questionnaire which measures adolescent health and functioning across education, legal, and family relations domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Stacy A Sterling, Oakland, California, United States

REFERENCES:
- [Background] Schmittdiel JA, Shortell SM, Rundall TG, Bodenheimer T, Selby JV. Effect of primary health care orientation on chronic care management. Ann Fam Med. 2006 Mar-Apr;4(2):117-23. doi: 10.1370/afm.520. PMID 16569714
- [Background] Selby JV, Uratsu CS, Fireman B, Schmittdiel JA, Peng T, Rodondi N, Karter AJ, Kerr EA. Treatment intensification and risk factor control: toward more clinically relevant quality measures. Med Care. 2009 Apr;47(4):395-402. doi: 10.1097/mlr.0b013e31818d775c. PMID 19330888
- [Background] Saunders KW, Davis RL, Stergachis A. Group Health Cooperative. In: Strom BL, ed. Pharmacoepidemiology. 4th ed. New York: Wiley, 2005:223-239
- [Background] Selby JV, Smith DH, Johnson ES, et al. Kaiser Permanente Medical Care Program. In: Strom BL, ed. Pharmacoepidemiology. 4th ed. New York: Wiley, 2005:241-259
- [Background] Babor TE, Higgins-Biddle J, Dauser D, Higgins P, Burleson JA. Alcohol screening and brief intervention in primary care settings: implementation models and predictors. J Stud Alcohol. 2005 May;66(3):361-8. doi: 10.15288/jsa.2005.66.361. PMID 16047525
- [Background] Brindis C, Park MJ, Ozer EM, Irwin CE Jr. Adolescents' access to health services and clinical preventive health care: crossing the great divide. Pediatr Ann. 2002 Sep;31(9):575-81. doi: 10.3928/0090-4481-20020901-10. No abstract available. PMID 12271742
- [Background] Blum R. Physicians' assessment of deficiencies and desire for training in adolescent care. J Med Educ. 1987 May;62(5):401-7. doi: 10.1097/00001888-198705000-00005. PMID 3573019
- [Background] Shrier LA, Harris SK, Kurland M, Knight JR. Substance use problems and associated psychiatric symptoms among adolescents in primary care. Pediatrics. 2003 Jun;111(6 Pt 1):e699-705. doi: 10.1542/peds.111.6.e699. PMID 12777588
- [Background] Cowell AJ, Bray JW, Mills MJ, Hinde JM. Conducting economic evaluations of screening and brief intervention for hazardous drinking: Methods and evidence to date for informing policy. Drug Alcohol Rev. 2010 Nov;29(6):623-30. doi: 10.1111/j.1465-3362.2010.00238.x. PMID 20973847
- [Background] Ockene JK, Adams A, Hurley TG, Wheeler EV, Hebert JR. Brief physician- and nurse practitioner-delivered counseling for high-risk drinkers: does it work? Arch Intern Med. 1999 Oct 11;159(18):2198-205. doi: 10.1001/archinte.159.18.2198. PMID 10527297
- [Background] Reiff-Hekking S, Ockene JK, Hurley TG, Reed GW. Brief physician and nurse practitioner-delivered counseling for high-risk drinking. Results at 12-month follow-up. J Gen Intern Med. 2005 Jan;20(1):7-13. doi: 10.1111/j.1525-1497.2005.21240.x. PMID 15693921
- [Background] McIntosh MC, Leigh G, Baldwin NJ, Marmulak J. Reducing alcohol consumption. Comparing three brief methods in family practice. Can Fam Physician. 1997 Nov;43:1959-62, 1965-7. PMID 9386883
- [Background] Babor TF, Higgins-Biddle JC, Dauser D, Burleson JA, Zarkin GA, Bray J. Brief interventions for at-risk drinking: patient outcomes and cost-effectiveness in managed care organizations. Alcohol Alcohol. 2006 Nov-Dec;41(6):624-31. doi: 10.1093/alcalc/agl078. Epub 2006 Oct 10. PMID 17035245
- [Background] Burke PJ, Da Silva JD, Vaughan BL, Knight JR. Training high school counselors on the use of motivational interviewing to screen for substance abuse. Subst Abus. 2005 Dec;26(3-4):31-4. doi: 10.1300/j465v26n03_07. PMID 16837410
- [Background] Goodall CA, Ayoub AF, Crawford A, Smith I, Bowman A, Koppel D, Gilchrist G. Nurse-delivered brief interventions for hazardous drinkers with alcohol-related facial trauma: a prospective randomised controlled trial. Br J Oral Maxillofac Surg. 2008 Mar;46(2):96-101. doi: 10.1016/j.bjoms.2007.11.014. Epub 2007 Dec 21. PMID 18160192
- [Background] Gil AG, Wagner EF, Tubman JG. Culturally sensitive substance abuse intervention for Hispanic and African American adolescents: empirical examples from the Alcohol Treatment Targeting Adolescents in Need (ATTAIN) Project. Addiction. 2004 Nov;99 Suppl 2:140-50. doi: 10.1111/j.1360-0443.2004.00861.x. PMID 15488112
- [Background] Grenard JL, Ames SL, Wiers RW, Thush C, Stacy AW, Sussman S. Brief intervention for substance use among at-risk adolescents: a pilot study. J Adolesc Health. 2007 Feb;40(2):188-91. doi: 10.1016/j.jadohealth.2006.08.008. Epub 2006 Oct 27. PMID 17259065
- [Background] Martin G, Copeland J, Swift W. The Adolescent Cannabis Check-Up: feasibility of a brief intervention for young cannabis users. J Subst Abuse Treat. 2005 Oct;29(3):207-13. doi: 10.1016/j.jsat.2005.06.005. PMID 16183469
- [Background] Winters KC, Leitten W, Wagner E, O'Leary Tevyaw T. Use of brief interventions for drug abusing teenagers within a middle and high school setting. J Sch Health. 2007 Apr;77(4):196-206. doi: 10.1111/j.1746-1561.2007.00191.x. PMID 17425522
- [Background] Srisurapanont M, Sombatmai S, Boripuntakul T. Brief intervention for students with methamphetamine use disorders: a randomized controlled trial. Am J Addict. 2007 Mar-Apr;16(2):111-6. doi: 10.1080/10550490601184431. PMID 17453612
- [Background] Suzuki K, Takeda A, Murakami S, Yuzuriha T, Hiezima M, Yoshimori C, Fuzibayashi T. [Brief intervention for smoking, problem drinking and drug abuse by high school students]. Nihon Arukoru Yakubutsu Igakkai Zasshi. 2003 Dec;38(6):475-82. Japanese. PMID 14750357
- [Background] Peterson PL, Baer JS, Wells EA, Ginzler JA, Garrett SB. Short-term effects of a brief motivational intervention to reduce alcohol and drug risk among homeless adolescents. Psychol Addict Behav. 2006 Sep;20(3):254-64. doi: 10.1037/0893-164X.20.3.254. PMID 16938063
- [Background] McCambridge J, Strang J. The efficacy of single-session motivational interviewing in reducing drug consumption and perceptions of drug-related risk and harm among young people: results from a multi-site cluster randomized trial. Addiction. 2004 Jan;99(1):39-52. doi: 10.1111/j.1360-0443.2004.00564.x. PMID 14678061
- [Background] Barroso T, Castanhola R, Marta M, et al. Effectiveness of brief alcohol interventions by clinical nurse specialists (CNS) in primary care settings. 2010 ISBRA World Congress, Paris, France, Sep 13-16, 2010
- [Background] National Institute on Alcohol Abuse and Alcoholism. Five-year strategic plan (FY07-11): Alcohol across the lifespan. Washington, DC: U.S. Department of Health and Human Services, 2006. http://pubs.niaaa.nih.gov/publications/StrategicPlan/NIAAASTRATEGICPLAN.htm. Accessed Oct 18, 2010.
- [Background] Institute of Medicine (US) Committee on Crossing the Quality Chasm: Adaptation to Mental Health and Addictive Disorders. Improving the Quality of Health Care for Mental and Substance-Use Conditions: Quality Chasm Series. Washington (DC): National Academies Press (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK19830/ PMID 20669433
- [Background] Chambers RA, Taylor JR, Potenza MN. Developmental neurocircuitry of motivation in adolescence: a critical period of addiction vulnerability. Am J Psychiatry. 2003 Jun;160(6):1041-52. doi: 10.1176/appi.ajp.160.6.1041. PMID 12777258
- [Background] Thatcher DL, Clark DB. Adolescents at risk for substance use disorders: role of psychological dysregulation, endophenotypes, and environmental influences. Alcohol Res Health. 2008;31(2):168-76. PMID 23584818
- [Background] Di Forti M, Morrison PD, Butt A, Murray RM. Cannabis use and psychiatric and cogitive disorders: the chicken or the egg? Curr Opin Psychiatry. 2007 May;20(3):228-34. doi: 10.1097/YCO.0b013e3280fa838e. PMID 17415074
- [Background] Ammon L, Sterling S, Mertens J, Weisner C. Adolescents in private chemical dependency programs: who are most at risk for HIV? J Subst Abuse Treat. 2005 Jul;29(1):39-45. doi: 10.1016/j.jsat.2005.03.003. PMID 15979530
- [Background] Substance Abuse and Mental Health Services Administration. SAMHSA Report to Congress - Nov 2002. The prevention and treatment of co-occurring substance abuse disorders and mental disorders. Rockville, MD, 2002. http://www.samhsa.gov/reports/congress2002/CoOccurringRpt.pdf. Accessed Oct 25, 2010
- [Background] Windle M, Spear LP, Fuligni AJ, Angold A, Brown JD, Pine D, Smith GT, Giedd J, Dahl RE. Transitions into underage and problem drinking: developmental processes and mechanisms between 10 and 15 years of age. Pediatrics. 2008 Apr;121 Suppl 4(Suppl 4):S273-89. doi: 10.1542/peds.2007-2243C. PMID 18381494
- [Background] Brown SA, Tapert SF, Granholm E, Delis DC. Neurocognitive functioning of adolescents: effects of protracted alcohol use. Alcohol Clin Exp Res. 2000 Feb;24(2):164-71. PMID 10698367
- [Background] Bava S, Tapert SF. Adolescent brain development and the risk for alcohol and other drug problems. Neuropsychol Rev. 2010 Dec;20(4):398-413. doi: 10.1007/s11065-010-9146-6. Epub 2010 Oct 19. PMID 20953990
- [Background] Kaplan JE, Benson C, Holmes KK, Brooks JT, Pau A, Masur H; Centers for Disease Control and Prevention (CDC); National Institutes of Health; HIV Medicine Association of the Infectious Diseases Society of America. Guidelines for prevention and treatment of opportunistic infections in HIV-infected adults and adolescents: recommendations from CDC, the National Institutes of Health, and the HIV Medicine Association of the Infectious Diseases Society of America. MMWR Recomm Rep. 2009 Apr 10;58(RR-4):1-207; quiz CE1-4. PMID 19357635
- [Background] Sisko AM, Truffer CJ, Keehan SP, Poisal JA, Clemens MK, Madison AJ. National health spending projections: the estimated impact of reform through 2019. Health Aff (Millwood). 2010 Oct;29(10):1933-41. doi: 10.1377/hlthaff.2010.0788. Epub 2010 Sep 9. PMID 20829295
- [Background] Mental Health America. Parity and health care reform: important changes for behavioral health, 2010. http://www.mentalhealthamerica.net/go/action/policy-issues-a-z/healthcare-reform. Accessed Oct 21, 2010
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Curley B. Healthcare reform law gives big boost to addiction treatment and prevention. Join Together. Apr 9, 2010. http://www.jointogether.org/news/features/2010/healthcare-reform-law-gives.html. Accessed Oct 21, 2010
- [Background] Johnston LD, O'Malley PM, Bachman JG, et al. Cigarette smoking among American teens continues to decline, but more slowly than in the past [press release]. Ann Arbor, MI: University of Michigan News and Information Services, 2006. http://www.monitoringthefuture.org/pressreleases/06cigpr.pdf. Accessed Oct 20, 2010
- [Background] National Institute on Alcohol Abuse and Alcoholism. Statistical snapshot of underage drinking, 2008. http://www.niaaa.nih.gov/AboutNIAAA/NIAAASponsoredPrograms/StatisticalSnapshotUnderageDrinking.htm. Accessed Oct 19, 2010
- [Background] Johnston LD, O'Malley PM, Bachman JG, et al. Monitoring the Future national results on adolescent drug use: Overview of key findings 2004. Bethesda, MD: National Institute on Drug Abuse, 2005. http://www.drugabuse.gov/PDF/overview2004.pdf. Accessed Oct 19, 2009
- [Background] Knight JR, Harris SK, Sherritt L, Van Hook S, Lawrence N, Brooks T, Carey P, Kossack R, Kulig J. Prevalence of positive substance abuse screen results among adolescent primary care patients. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1035-41. doi: 10.1001/archpedi.161.11.1035. PMID 17984404
- [Background] Underage Drinking Enforcement Training Center. Welcome to the Underage Drinking Enforcement Training Center. http://www.udetc.org/index.asp. Updated Oct 2010. Accessed Oct 27, 2010
- [Background] Office of National Drug Control Policy. The economic costs of drug abuse in the United States, 1992-2002. Washington, DC: Executive Office of the President (Publication No. 207303), 2004
- [Background] Merenstein D, Green L, Fryer GE, Dovey S. Shortchanging adolescents: room for improvement in preventive care by physicians. Fam Med. 2001 Feb;33(2):120-3. PMID 11271739
- [Background] Levy S, Vaughan BL, Knight JR. Office-based intervention for adolescent substance abuse. Pediatr Clin North Am. 2002 Apr;49(2):329-43. doi: 10.1016/s0031-3955(01)00007-4. PMID 11993286
- [Background] Yoast RA, Fleming M, Balch GI. Reactions to a concept for physician intervention in adolescent alcohol use. J Adolesc Health. 2007 Jul;41(1):35-41. doi: 10.1016/j.jadohealth.2007.02.008. Epub 2007 May 3. PMID 17577532
- [Background] Brown JD, Wissow LS. Discussion of sensitive health topics with youth during primary care visits: relationship to youth perceptions of care. J Adolesc Health. 2009 Jan;44(1):48-54. doi: 10.1016/j.jadohealth.2008.06.018. Epub 2008 Oct 25. PMID 19101458
- [Background] Sterling S, Weisner C. The role of primary care in addressing adolescent substance use: Screening, treatment, and coordination. Paper presented at the
- [Background] Kaul P, Coupey SM. Clinical evaluation of substance abuse. Pediatr Rev. 2002 Mar;23(3):85-94. doi: 10.1542/pir.23-3-85. No abstract available. PMID 11875181
- [Background] Knight JR. The role of the primary care provider in preventing and treating alcohol problems in adolescents. Ambul Pediatr. 2001 May-Jun;1(3):150-61. doi: 10.1367/1539-4409(2001)0012.0.co;2. PMID 11888392
- [Background] Indications for management and referral of patients involved in substance abuse. American Academy of Pediatrics. Committee on Substance Abuse. Pediatrics. 2000 Jul;106(1 Pt 1):143-8. doi: 10.1542/peds.106.1.143. PMID 10878166
- [Background] American Academy of Pediatrics. Committee on Substance Abuse. American Academy of Pediatrics. Committee on Substance Abuse. Tobacco, alcohol, and other drugs: the role of the pediatrician in prevention and management of substance abuse. Pediatrics. 1998 Jan;101(1 Pt 1):125-8. PMID 11345974
- [Background] Elster A. The American Medical Association Guidelines for Adolescent Preventive Services. Arch Pediatr Adolesc Med. 1997 Sep;151(9):958-9. doi: 10.1001/archpedi.1997.02170460096021. No abstract available. PMID 9308880
- [Background] U.S. Preventive Services Task Force. The Guide to Clinical Preventive Services 2010 - 2011: Recommendations of the U.S. Preventive Services Task Force. Rockville (MD): Agency for Healthcare Research and Quality (US); 2010 Aug. Report No.: 10-05145. Available from http://www.ncbi.nlm.nih.gov/books/NBK56707/ PMID 21850778
- [Background] American Academy of Pediatrics. Periodic survey of fellows: 45% of Fellows routinely screen for alcohol use., 2002. http://aapnews.aappublications.org/cgi/content/short/14/10/1. Accessed April 6, 2009
- [Background] Bethell C, Klein J, Peck C. Assessing health system provision of adolescent preventive services: the Young Adult Health Care Survey. Med Care. 2001 May;39(5):478-90. doi: 10.1097/00005650-200105000-00008. PMID 11317096
- [Background] Friedman LS, Johnson B, Brett AS. Evaluation of substance-abusing adolescents by primary care physicians. J Adolesc Health Care. 1990 May;11(3):227-30. doi: 10.1016/0197-0070(90)90353-4. PMID 2358391
- [Background] Wilson CR, Sherritt L, Gates E, Knight JR. Are clinical impressions of adolescent substance use accurate? Pediatrics. 2004 Nov;114(5):e536-40. doi: 10.1542/peds.2004-0098. PMID 15520086
- [Background] Emans SJ, Bravender T, Knight J, Frazer C, Luoni M, Berkowitz C, Armstrong E, Goodman E. Adolescent medicine training in pediatric residency programs: are we doing a good job? Pediatrics. 1998 Sep;102(3 Pt 1):588-95. doi: 10.1542/peds.102.3.588. PMID 9738181
- [Background] Leontieva L, Horn K, Haque A, Helmkamp J, Ehrlich P, Williams J. Readiness to change problematic drinking assessed in the emergency department as a predictor of change. J Crit Care. 2005 Sep;20(3):251-6. doi: 10.1016/j.jcrc.2005.05.009. PMID 16253794
- [Background] Lawendowski LA. A motivational intervention for adolescent smokers. Prev Med. 1998 Sep-Oct;27(5 Pt 3):A39-46. doi: 10.1006/pmed.1998.0424. PMID 9808816
- [Background] Knight JR, Sherritt L, Van Hook S, Gates EC, Levy S, Chang G. Motivational interviewing for adolescent substance use: a pilot study. J Adolesc Health. 2005 Aug;37(2):167-9. doi: 10.1016/j.jadohealth.2004.08.020. PMID 16026730
- [Background] Marlatt GA, Baer JS, Kivlahan DR, Dimeff LA, Larimer ME, Quigley LA, Somers JM, Williams E. Screening and brief intervention for high-risk college student drinkers: results from a 2-year follow-up assessment. J Consult Clin Psychol. 1998 Aug;66(4):604-15. doi: 10.1037//0022-006x.66.4.604. PMID 9735576
- [Background] Baer JS, Kivlahan DR, Blume AW, McKnight P, Marlatt GA. Brief intervention for heavy-drinking college students: 4-year follow-up and natural history. Am J Public Health. 2001 Aug;91(8):1310-6. doi: 10.2105/ajph.91.8.1310. PMID 11499124
- [Background] Borsari B, Carey KB. Effects of a brief motivational intervention with college student drinkers. J Consult Clin Psychol. 2000 Aug;68(4):728-33. PMID 10965648
- [Background] Carey KB, Correia CJ. Drinking motives predict alcohol-related problems in college students. J Stud Alcohol. 1997 Jan;58(1):100-5. doi: 10.15288/jsa.1997.58.100. PMID 8979218
- [Background] Barnett NP, Monti PM, Wood MD. Motivational interviewing for alcohol-involved adolescents in the emergency room. . In: Wagner EF, Waldron HB, eds. Innovations in Adolescent Substance Abuse Interventions. Amsterdam, Netherlands: Pergamon/Elsevier Science Inc, 2001:143-168
- [Background] Larimer ME, Turner AP, Anderson BK, Fader JS, Kilmer JR, Palmer RS, Cronce JM. Evaluating a brief alcohol intervention with fraternities. J Stud Alcohol. 2001 May;62(3):370-80. doi: 10.15288/jsa.2001.62.370. PMID 11414347
- [Background] Murphy JG, Duchnick JJ, Vuchinich RE, Davison JW, Karg RS, Olson AM, Smith AF, Coffey TT. Relative efficacy of a brief motivational intervention for college student drinkers. Psychol Addict Behav. 2001 Dec;15(4):373-9. doi: 10.1037//0893-164x.15.4.373. PMID 11767271
- [Background] Spirito A, Monti PM, Barnett NP, Colby SM, Sindelar H, Rohsenow DJ, Lewander W, Myers M. A randomized clinical trial of a brief motivational intervention for alcohol-positive adolescents treated in an emergency department. J Pediatr. 2004 Sep;145(3):396-402. doi: 10.1016/j.jpeds.2004.04.057. PMID 15343198
- [Background] Monti PM, Colby SM, Barnett NP, Spirito A, Rohsenow DJ, Myers M, Woolard R, Lewander W. Brief intervention for harm reduction with alcohol-positive older adolescents in a hospital emergency department. J Consult Clin Psychol. 1999 Dec;67(6):989-94. doi: 10.1037//0022-006x.67.6.989. PMID 10596521
- [Background] Tait RJ, Hulse GK, Robertson SI, Sprivulis PC. Emergency department-based intervention with adolescent substance users: 12-month outcomes. Drug Alcohol Depend. 2005 Sep 1;79(3):359-63. doi: 10.1016/j.drugalcdep.2005.03.015. Epub 2005 Apr 26. PMID 16102378
- [Background] D'Amico EJ, Miles JN, Stern SA, Meredith LS. Brief motivational interviewing for teens at risk of substance use consequences: a randomized pilot study in a primary care clinic. J Subst Abuse Treat. 2008 Jul;35(1):53-61. doi: 10.1016/j.jsat.2007.08.008. Epub 2007 Nov 26. PMID 18037603
- [Background] Gates S, McCambridge J, Smith LA, Foxcroft DR. Interventions for prevention of drug use by young people delivered in non-school settings. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005030. doi: 10.1002/14651858.CD005030.pub2. PMID 16437511
- [Background] Ozer EM, Adams SH, Lustig JL, Millstein SG, Camfield K, El-Diwany S, Volpe S, Irwin CE Jr. Can it be done? Implementing adolescent clinical preventive services. Health Serv Res. 2001 Dec;36(6 Pt 2):150-65. PMID 16148966
- [Background] Bien TH, Miller WR, Tonigan JS. Brief interventions for alcohol problems: a review. Addiction. 1993 Mar;88(3):315-35. doi: 10.1111/j.1360-0443.1993.tb00820.x. PMID 8461850
- [Background] D'Onofrio G, Degutis LC. Preventive care in the emergency department: screening and brief intervention for alcohol problems in the emergency department: a systematic review. Acad Emerg Med. 2002 Jun;9(6):627-38. doi: 10.1111/j.1553-2712.2002.tb02304.x. PMID 12045080
- [Background] Kanouse DE, Kallich JD, Kahan JP. Dissemination of effectiveness and outcomes research. Health Policy. 1995 Dec;34(3):167-92. doi: 10.1016/0168-8510(95)00760-1. PMID 10153899
- [Background] Bertholet N, Daeppen JB, Wietlisbach V, Fleming M, Burnand B. Reduction of alcohol consumption by brief alcohol intervention in primary care: systematic review and meta-analysis. Arch Intern Med. 2005 May 9;165(9):986-95. doi: 10.1001/archinte.165.9.986. PMID 15883236
- [Background] Kaner E, Bland M, Cassidy P, et al. Screening and brief alcohol intervention in routine primary care In the UK: SIPS trial outcomes at six months. 2010 ISBRA World Congress, Paris, France, Sep 13-16, 2010
- [Background] Clark DB, Gordon AJ, Ettaro LR, Owens JM, Moss HB. Screening and brief intervention for underage drinkers. Mayo Clin Proc. 2010 Apr;85(4):380-91. doi: 10.4065/mcp.2008.0638. PMID 20360296
- [Background] Friedmann PD, McCullough D, Saitz R. Screening and intervention for illicit drug abuse: a national survey of primary care physicians and psychiatrists. Arch Intern Med. 2001 Jan 22;161(2):248-51. doi: 10.1001/archinte.161.2.248. PMID 11176739
- [Background] Ewing GB, Selassie AW, Lopez CH, McCutcheon EP. Self-report of delivery of clinical preventive services by U.S. physicians. Comparing specialty, gender, age, setting of practice, and area of practice. Am J Prev Med. 1999 Jul;17(1):62-72. doi: 10.1016/s0749-3797(99)00032-x. PMID 10429755
- [Background] Klein JD, Wilson KM. Delivering quality care: adolescents' discussion of health risks with their providers. J Adolesc Health. 2002 Mar;30(3):190-5. doi: 10.1016/s1054-139x(01)00342-1. PMID 11869926
- [Background] Mertens JR, Flisher AJ, Fleming MF, Weisner CM. Medical conditions of adolescents in alcohol and drug treatment: comparison with matched controls. J Adolesc Health. 2007 Feb;40(2):173-9. doi: 10.1016/j.jadohealth.2006.09.021. Epub 2006 Nov 29. PMID 17259058
- [Background] Sterling S, Kohn C, Lu Y, Weisner C. Pathways to chemical dependency treatment for adolescents in an HMO. J Psychoactive Drugs. 2004 Dec;36(4):439-53. doi: 10.1080/02791072.2004.10524427. PMID 15751482
- [Background] Saitz R, Svikis D, D'Onofrio G, Kraemer KL, Perl H. Challenges applying alcohol brief intervention in diverse practice settings: populations, outcomes, and costs. Alcohol Clin Exp Res. 2006 Feb;30(2):332-8. doi: 10.1111/j.1530-0277.2006.00038.x. PMID 16441282
- [Background] Massachusetts Department of Public Health Bureau of Substance Abuse Services. Provider Guide: Adolescent Screening, Brief Intervention, and Referral to Treatment Using the CRAFFT Screening Tool. Boston: Massachusetts Department of Public Health, 2009
- [Background] Phillips JL, Smithstan P. Brief intervention: An approach for substance abusing adolescents. Trainer and trainee guide. A CARS training program prepared by Joel L. Phillips and Pam Smithstan, MFT, based on the work of Ken Winters, PhD. Santa Rosa, CA: Center for Applied Research Solutions, 2006. http://indianeducation.org/userfiles/file/Session%207_3b%20Brief%20Intervention%20FBecker.pdf
- [Background] Barry KL, Blow FC, Willenbring ML, McCormick R, Brockmann LM, Visnic S. Use of Alcohol Screening and Brief Interventions<br />in Primary Care Settings:Implementation and Barriers. Subst Abus. 2004 Mar;25(1):27-36. doi: 10.1300/J465v25n01_05. PMID 15201109
- [Background] Friedmann PD, McCullough D, Chin MH, Saitz R. Screening and intervention for alcohol problems. A national survey of primary care physicians and psychiatrists. J Gen Intern Med. 2000 Feb;15(2):84-91. doi: 10.1046/j.1525-1497.2000.03379.x. PMID 10672110
- [Background] Spandorfer JM, Israel Y, Turner BJ. Primary care physicians' views on screening and management of alcohol abuse: inconsistencies with national guidelines. J Fam Pract. 1999 Nov;48(11):899-902. PMID 10907628
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Background] Gottlieb NH, Mullen PD, McAlister AL. Patients' substance abuse and the primary care physician: patterns of practice. Addict Behav. 1987;12(1):23-32. doi: 10.1016/0306-4603(87)90005-0. PMID 3565109
- [Background] Miller NS, Sheppard LM, Colenda CC, Magen J. Why physicians are unprepared to treat patients who have alcohol- and drug-related disorders. Acad Med. 2001 May;76(5):410-8. doi: 10.1097/00001888-200105000-00007. PMID 11346513
- [Background] Ogborne AC, Rush B, Ekdahl A, Fondacaro R. The views of health and social service professionals regarding alcohol problems and their treatment. Int J Addict. 1986 Sep-Oct;21(9-10):1051-8. doi: 10.3109/10826088609077254. PMID 3793309
- [Background] Ozer EM, Adams SH, Gardner LR, Mailloux DE, Wibbelsman CJ, Irwin CE Jr. Provider self-efficacy and the screening of adolescents for risky health behaviors. J Adolesc Health. 2004 Aug;35(2):101-7. doi: 10.1016/j.jadohealth.2003.09.016. PMID 15261638
- [Background] Saitz R, Friedmann PD, Sullivan LM, Winter MR, Lloyd-Travaglini C, Moskowitz MA, Samet JH. Professional satisfaction experienced when caring for substance-abusing patients: faculty and resident physician perspectives. J Gen Intern Med. 2002 May;17(5):373-6. doi: 10.1046/j.1525-1497.2002.10520.x. PMID 12047735
- [Background] Westermeyer J, Doheny S, Stone B. An assessment of hospital care for the alcoholic patient. Alcohol Clin Exp Res. 1978 Jan;2(1):53-7. doi: 10.1111/j.1530-0277.1978.tb04694.x. PMID 345854
- [Background] Gardner W, Pajer KA, Kelleher KJ, Scholle SH, Wasserman RC. Child sex differences in primary care clinicians' mental health care of children and adolescents. Arch Pediatr Adolesc Med. 2002 May;156(5):454-9. doi: 10.1001/archpedi.156.5.454. PMID 11980550
- [Background] Gardner W, Kelleher KJ, Pajer KA, Campo JV. Primary care clinicians' use of standardized tools to assess child psychosocial problems. Ambul Pediatr. 2003 Jul-Aug;3(4):191-5. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 12882596
- [Background] Volk RJ, Steinbauer JR, Cantor SB. Patient factors influencing variation in the use of preventive interventions for alcohol abuse by primary care physicians. J Stud Alcohol. 1996 Mar;57(2):203-9. doi: 10.15288/jsa.1996.57.203. PMID 8683970
- [Background] McCrady BS, Richter SS, Morgan TJ, Slade J, Pfeifer C. Involving health care workers in screening for alcohol problems. J Addict Dis. 1996;15(3):45-58. doi: 10.1300/J069v15n03_03. PMID 8842849
- [Background] Franzgrote M, Ellen JM, Millstein SG, Irwin CE Jr. Screening for adolescent smoking among primary care physicians in California. Am J Public Health. 1997 Aug;87(8):1341-5. doi: 10.2105/ajph.87.8.1341. PMID 9279272
- [Background] Ellen JM, Franzgrote M, Irwin CE Jr, Millstein SG. Primary care physicians' screening of adolescent patients: a survey of California physicians. J Adolesc Health. 1998 Jun;22(6):433-8. doi: 10.1016/s1054-139x(97)00276-0. PMID 9627812
- [Background] Barnett NP, Monti PM, Cherpitel C, Bendtsen P, Borges G, Colby SM, Nordqvist C, Johansson K. Identification and brief treatment of alcohol problems with medical patients: an international perspective. Alcohol Clin Exp Res. 2003 Feb;27(2):262-70. doi: 10.1097/01.ALC.0000057123.36127.8B. PMID 12605075
- [Background] Sterling S, Weisner C, Hinman A, Parthasarathy S. Access to treatment for adolescents with substance use and co-occurring disorders: challenges and opportunities. J Am Acad Child Adolesc Psychiatry. 2010 Jul;49(7):637-46; quiz 725-6. doi: 10.1016/j.jaac.2010.03.019. Epub 2010 May 8. PMID 20610133
- [Background] Parthasarathy S, Weisner C. Health care services use by adolescents with intakes into an outpatient alcohol and drug treatment program. Am J Addict. 2006;15 Suppl 1:113-21. doi: 10.1080/10550490601006097. PMID 17182426
- [Background] Sterling S, Weisner C. Chemical dependency and psychiatric services for adolescents in private managed care: implications for outcomes. Alcohol Clin Exp Res. 2005 May;29(5):801-9. doi: 10.1097/01.alc.0000164373.89061.2c. PMID 15897726
- [Background] Sterling S, Weisner C. Translating research findings into practice: example of treatment services for adolescents in managed care. Alcohol Res Health. 2006;29(1):11-8. PMID 16767848
- [Background] Sterling S, Chi F, Campbell C, Weisner C. Three-year chemical dependency and mental health treatment outcomes among adolescents: the role of continuing care. Alcohol Clin Exp Res. 2009 Aug;33(8):1417-29. doi: 10.1111/j.1530-0277.2009.00972.x. Epub 2009 Apr 30. PMID 19413644
- [Background] Wu NS, Lu Y, Sterling S, Weisner C. Family environment factors and substance abuse severity in an HMO adolescent treatment population. Clin Pediatr (Phila). 2004 May;43(4):323-33. doi: 10.1177/000992280404300403. PMID 15118775
- [Background] Campbell CI, Chi F, Sterling S, Kohn C, Weisner C. Self-initiated tobacco cessation and substance use outcomes among adolescents entering substance use treatment in a managed care organization. Addict Behav. 2009 Feb;34(2):171-9. doi: 10.1016/j.addbeh.2008.10.002. Epub 2008 Oct 10. PMID 19010600
- [Background] Chi FW, Sterling S, Campbell CI, et al. Twelve-step participation at 5-year follow-up among a diverse sample of adolescents entering chemical dependency treatment. Joint Meeting on Adolescent Treatment Effectiveness (JMATE), Washington, DC, Mar 25-27, 2008
- [Background] Scott M, Parthasarathy S, Kohn C, Hinman A, Sterling S, Weisner C. Adolescents with substance diagnoses in an HMO: factors associated with medical provider referrals to substance abuse and mental health treatment. Ment Health Serv Res. 2004 Mar;6(1):47-60. doi: 10.1023/b:mhsr.0000011256.70502.ed. PMID 15002680
- [Background] Chi FW, Sterling S, Weisner C. Adolescents with co-occurring substance use and mental conditions in a private managed care health plan: prevalence, patient characteristics, and treatment initiation and engagement. Am J Addict. 2006;15 Suppl 1:67-79. doi: 10.1080/10550490601006022. PMID 17182422
- [Background] Mertens JR, Weisner C, Ray GT, Fireman B, Walsh K. Hazardous drinkers and drug users in HMO primary care: prevalence, medical conditions, and costs. Alcohol Clin Exp Res. 2005 Jun;29(6):989-98. doi: 10.1097/01.alc.0000167958.68586.3d. PMID 15976525
- [Background] Mertens JR, Lu YW, Parthasarathy S, Moore C, Weisner CM. Medical and psychiatric conditions of alcohol and drug treatment patients in an HMO: comparison with matched controls. Arch Intern Med. 2003 Nov 10;163(20):2511-7. doi: 10.1001/archinte.163.20.2511. PMID 14609789
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Lu Y. Integrating primary medical care with addiction treatment: a randomized controlled trial. JAMA. 2001 Oct 10;286(14):1715-23. doi: 10.1001/jama.286.14.1715. PMID 11594896
- [Background] Chi FW, Weisner CM. Nine-year psychiatric trajectories and substance use outcomes: an application of the group-based modeling approach. Eval Rev. 2008 Feb;32(1):39-58. doi: 10.1177/0193841X07307317. PMID 18198170
- [Background] Parthasarathy S, Weisner C, Hu TW, Moore C. Association of outpatient alcohol and drug treatment with health care utilization and cost: revisiting the offset hypothesis. J Stud Alcohol. 2001 Jan;62(1):89-97. doi: 10.15288/jsa.2001.62.89. PMID 11271969
- [Background] Parthasarathy S, Weisner CM. Five-year trajectories of health care utilization and cost in a drug and alcohol treatment sample. Drug Alcohol Depend. 2005 Nov 1;80(2):231-40. doi: 10.1016/j.drugalcdep.2005.04.004. PMID 15916868
- [Background] Alexandre PK, French MT, Matzger H, Weisner C. Addiction treatment history, medical services utilization, and cost: a longitudinal analysis of problem drinkers. J Addict Dis. 2006;25(1):105-20. doi: 10.1300/J069v25n01_13. PMID 16597578
- [Background] Van Den Eeden SK, Tanner CM, Bernstein AL, Fross RD, Leimpeter A, Bloch DA, Nelson LM. Incidence of Parkinson's disease: variation by age, gender, and race/ethnicity. Am J Epidemiol. 2003 Jun 1;157(11):1015-22. doi: 10.1093/aje/kwg068. PMID 12777365
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- [Background] Knight JR, Sherritt L, Harris SK, Gates EC, Chang G. Validity of brief alcohol screening tests among adolescents: a comparison of the AUDIT, POSIT, CAGE, and CRAFFT. Alcohol Clin Exp Res. 2003 Jan;27(1):67-73. doi: 10.1097/01.ALC.0000046598.59317.3A. PMID 12544008
- [Background] Wibbelsman CJ. Confidentiality in an Age of Managed Care: Can It Exist? Adolesc Med. 1997 Oct;8(3):427-432. PMID 10360023
- [Background] Desy PM, Perhats C. Alcohol screening, brief intervention, and referral in the emergency department: an implementation study. J Emerg Nurs. 2008 Feb;34(1):11-9. doi: 10.1016/j.jen.2007.03.019. Epub 2007 Dec 3. PMID 18237661
- [Background] Fleming MF. Strategies to increase alcohol screening in health care settings. Alcohol Health Res World. 1997;21(4):340-7. PMID 15706746
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People for Change. 2nd ed. New York: Guilford Press, 2002
- [Background] Moyers TB, Martin T, Manuel JK, Hendrickson SM, Miller WR. Assessing competence in the use of motivational interviewing. J Subst Abuse Treat. 2005 Jan;28(1):19-26. doi: 10.1016/j.jsat.2004.11.001. PMID 15723728
- [Background] Hunkeler EM, Meresman JF, Hargreaves WA, Fireman B, Berman WH, Kirsch AJ, Groebe J, Hurt SW, Braden P, Getzell M, Feigenbaum PA, Peng T, Salzer M. Efficacy of nurse telehealth care and peer support in augmenting treatment of depression in primary care. Arch Fam Med. 2000 Aug;9(8):700-8. doi: 10.1001/archfami.9.8.700. PMID 10927707
- [Background] Meresman JF, Hunkeler EM, Hargreaves WA, Kirsch AJ, Robinson P, Green A, Mann EZ, Getzell M, Feigenbaum P. A case report: implementing a nurse telecare program for treating depression in primary care. Psychiatr Q. 2003 Spring;74(1):61-73. doi: 10.1023/a:1021145722959. PMID 12602789
- [Background] Fraser D. The depression initiative: an alliance to improve treatment. The Permanente Journal. 1998;2 (3):5-11
- [Background] Aspy CB, Mold JW, Thompson DM, Blondell RD, Landers PS, Reilly KE, Wright-Eakers L. Integrating screening and interventions for unhealthy behaviors into primary care practices. Am J Prev Med. 2008 Nov;35(5 Suppl):S373-80. doi: 10.1016/j.amepre.2008.08.015. PMID 18929984
- [Background] Leffingwell TR. Motivational Interviewing Knowledge and Attitudes Test (MIKAT) for evaluation of training outcomes. Minuet. 2006;13 (1):10-11
- [Background] Meyers K, McLellan AT, Jaeger JL, Pettinati HM. The development of the Comprehensive Addiction Severity Index for Adolescents (CASI-A). An interview for assessing multiple problems of adolescents. J Subst Abuse Treat. 1995 May-Jun;12(3):181-93. doi: 10.1016/0740-5472(95)00009-t. PMID 7474026
- [Background] Whitmore EA, Mikulich SK, Thompson LL, Riggs PD, Aarons GA, Crowley TJ. Influences on adolescent substance dependence: conduct disorder, depression, attention deficit hyperactivity disorder, and gender. Drug Alcohol Depend. 1997 Aug 25;47(2):87-97. doi: 10.1016/s0376-8716(97)00074-4. PMID 9298330
- [Background] Ammon L, Lu Y, Weisner C. Adolescents in substance abuse treatment: Are they at risk for HIV? 131st meeting of American Public Health Association, San Francisco, CA, 2003
- [Background] Balsa AI, Homer JF, French MT, Weisner CM. Substance use, education, employment, and criminal activity outcomes of adolescents in outpatient chemical dependency programs. J Behav Health Serv Res. 2009 Jan;36(1):75-95. doi: 10.1007/s11414-007-9095-x. Epub 2007 Dec 7. PMID 18064572
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Hunkeler EM, Hu T, Selby JV. The outcome and cost of alcohol and drug treatment in an HMO: day hospital versus traditional outpatient regimens. Health Serv Res. 2000 Oct;35(4):791-812. PMID 11055449
- [Background] Parthasarathy S, Mertens J, Moore C, Weisner C. Utilization and cost impact of integrating substance abuse treatment and primary care. Med Care. 2003 Mar;41(3):357-67. doi: 10.1097/01.MLR.0000053018.20700.56. PMID 12618639
- [Background] Hsiao C. Analysis of Panel Data. New York: Cambridge University Press, 1986
- [Background] Muthén B, Kaplan D, Hollis M. On structural equation modeling with data that are not missing completely at random. Psychometrika. 1987;42:431-462
- [Background] Sterling S, Weisner C. Improving retention among women in substance abuse treatment: Is childcare enough? 129th meeting of the American Public Health Association, Atlanta, GA, 2001
- [Background] Qualitative Solutions and Research: QSR NUD*IST [computer program]. 5.0. Thousand Oaks, CA: Sage Publications; 2000
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. Hillsdale, NJ: Lawrence Erlbaum Associates, Inc., 1988
- [Background] Killip S, Mahfoud Z, Pearce K. What is an intracluster correlation coefficient? Crucial concepts for primary care researchers. Ann Fam Med. 2004 May-Jun;2(3):204-8. doi: 10.1370/afm.141. PMID 15209195
- [Background] de Leeuw J, Kreft IG. Questioning multilevel models. J Educ Behav Stat. 1995;20 (2):171-189
- [Background] Bryk AS, Raudenbush SW. Hierarchical Linear Models: Applications and Data Analysis Methods. Newbury Park: Sage, 1992
- [Background] Barrientos-Gutierrez T, Gimeno D, Mangione TW, Harrist RB, Amick BC. Drinking social norms and drinking behaviours: a multilevel analysis of 137 workgroups in 16 worksites. Occup Environ Med. 2007 Sep;64(9):602-8. doi: 10.1136/oem.2006.031765. Epub 2007 May 24. PMID 17525095
- [Background] Cosby RH, Howard M, Kaczorowski J, Willan AR, Sellors JW. Randomizing patients by family practice: sample size estimation, intracluster correlation and data analysis. Fam Pract. 2003 Feb;20(1):77-82. doi: 10.1093/fampra/20.1.77. PMID 12509376
- [Background] Slymen DJ, Hovell MF. Cluster versus individual randomization in adolescent tobacco and alcohol studies: illustrations for design decisions. Int J Epidemiol. 1997 Aug;26(4):765-71. doi: 10.1093/ije/26.4.765. PMID 9279608
- [Background] Mertens JR, Flisher AJ, Satre DD, Weisner CM. The role of medical conditions and primary care services in 5-year substance use outcomes among chemical dependency treatment patients. Drug Alcohol Depend. 2008 Nov 1;98(1-2):45-53. doi: 10.1016/j.drugalcdep.2008.04.007. Epub 2008 Jun 20. PMID 18571875
- [Background] Mertens JR, Weisner CM. Predictors of substance abuse treatment retention among women and men in an HMO. Alcohol Clin Exp Res. 2000 Oct;24(10):1525-33. PMID 11045861
- [Background] Weisner C, Delucchi K, Matzger H, Schmidt L. The role of community services and informal support on five-year drinking trajectories of alcohol dependent and problem drinkers. J Stud Alcohol. 2003 Nov;64(6):862-73. doi: 10.15288/jsa.2003.64.862. PMID 14743951
- [Background] Weisner C, Matzger H. Missed opportunities in addressing drinking behavior in medical and mental health services. Alcohol Clin Exp Res. 2003 Jul;27(7):1132-41. doi: 10.1097/01.ALC.0000075546.38349.69. PMID 12878919
- [Background] Weisner C, Schmidt LA. Rethinking access to alcohol treatment. Recent Dev Alcohol. 2001;15:107-36. doi: 10.1007/978-0-306-47193-3_7. No abstract available. PMID 11449738
- [Derived] Sterling S, Parthasarathy S, Jones A, Weisner C, Metz V, Hartman L, Saba K, Kline-Simon AH. Young Adult Substance Use and Healthcare Use Associated With Screening, Brief Intervention and Referral to Treatment in Pediatric Primary Care. J Adolesc Health. 2022 Oct;71(4S):S15-S23. doi: 10.1016/j.jadohealth.2021.11.033. PMID 36122965
- [Derived] Parthasarathy S, Kline-Simon AH, Jones A, Hartman L, Saba K, Weisner C, Sterling S. Three-Year Outcomes After Brief Treatment of Substance Use and Mood Symptoms. Pediatrics. 2021 Jan;147(1):e2020009191. doi: 10.1542/peds.2020-009191. PMID 33372122
- [Derived] Sterling S, Kline-Simon AH, Weisner C, Jones A, Satre DD. Pediatrician and Behavioral Clinician-Delivered Screening, Brief Intervention and Referral to Treatment: Substance Use and Depression Outcomes. J Adolesc Health. 2018 Apr;62(4):390-396. doi: 10.1016/j.jadohealth.2017.10.016. Epub 2018 Feb 1. PMID 29396080
- [Derived] Sterling S, Kline-Simon AH, Jones A, Satre DD, Parthasarathy S, Weisner C. Specialty addiction and psychiatry treatment initiation and engagement: Results from an SBIRT randomized trial in pediatrics. J Subst Abuse Treat. 2017 Nov;82:48-54. doi: 10.1016/j.jsat.2017.09.005. Epub 2017 Sep 10. PMID 29021115
- [Derived] Sterling S, Kline-Simon AH, Satre DD, Jones A, Mertens J, Wong A, Weisner C. Implementation of Screening, Brief Intervention, and Referral to Treatment for Adolescents in Pediatric Primary Care: A Cluster Randomized Trial. JAMA Pediatr. 2015 Nov;169(11):e153145. doi: 10.1001/jamapediatrics.2015.3145. Epub 2015 Nov 2. PMID 26523821